CLINICAL TRIAL: NCT04552002
Title: The Effect of Synbiotic Consumption on Glycemic, Inflammatory Markers and Body Composition on Prediabetic and Diabetic Patients: A Double Blinded Randomized Control Trial
Brief Title: The Effect of Synbiotic Consumption on Glycemic, Inflammatory Markers and Body Composition on Prediabetic and Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Razan Algarni, Principal investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2019-03-227
Record Dates: First submitted 2020-09-01; First posted 2020-09-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic group (Experimental): Intervention group:
  Will receive synbiotic supplements: one capsule/day. Each capsule contains 20 billion CFU multi-strain probiotics + prebiotics (inulin and oligosaccharides) for a duration of 6 months.
  Interventions: Dietary Supplement: Synbiotic group
- Placebo group (No Intervention): Will receive a placebo. The placebo will be similar to the synbiotic supplements in appearance.

INTERVENTIONS:
Dietary Supplement: Synbiotic group — Probiotics and prebiotics
  Arms: Synbiotic group

SUMMARY:
This is a randomized controlled trial that will be conducted on Saudi prediabetic and diabetic adults aged 18 to 70 years. The aim of the study is to investigate the effect of synbiotic consumption on gut microbiome, glycemic control, and other diabetes-related outcomes in patients with prediabetes and diabetes. A total of 160 participants will be recruited from King Fahd Hospital of the University, Eastern Province, Saudi Arabia and randomly assigned to synbiotic group (prediabetic and diabetic, n=40 each group) or control group (prediabetic and diabetic, n=40 each group) for a 6-month trial. A structured questionnaire will be used for data collection from subjects. The questionnaire will include data related to socioeconomic status, health and diet related history. Primary outcomes including gut microbiome sequencing, glycemic control related parameters and secondary outcomes including inflammatory markers, food intolerance and anthropometric measurements will be measured before the study, after 3 months and after 6 months. The findings of the current study will shed light on the significance of synbiotic consumption on glycemic control and other diabetes-related outcomes and their relation to food allergy and autoimmunity.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 1 diabetes
* Patients on insulin therapy
* Patients on antibiotics
* Pregnant and lactating women
* Smoking individuals
* Patients with comorbidities (except for hyperlipidemia and blood pressure)
* Patients taking immunosuppressants
* Patients taking probiotics, prebiotics or synbiotics

Exclusion Criteria:

* Patients with prediabetes (HbA1c of 5.7- 6.4% or a fasting plasma glucose of 100 -125 mg/dl)
* Patients with type 2 diabetes (HbA1c of ≥ 6.5% or a fasting plasma glucose of ≥ 126 mg/dl
* Male and female patients aged (18-70) years
* Patients with HbA1c of ≥ 5.7 or a fasting plasma glucose of ≥100 mg/dl
* BMI ≥ 25

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Glycemic markers | 6 months
  HbA1c, FBG (through blood samples)
Inflammatory markers | 6 months
  IL-1, IL-10, CRP, IFN-γ (through blood samples)
Body Composition parameters | 6 months
  Muscle mass, Fat mass (through a body composition analyzer)
BMI | 6 months
  Height and weight will be measured to obtain BMI (kg/m2)
Waist circumference | 6 months
  in (cm) by a measurement tape

SECONDARY OUTCOMES:
Microbiome sequencing | 6 months
  Will be obtained through stool samples

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Family Medicince Community Centre, Dammam, Eastern Province
  - King Fahd University Hospital, Dammam, Eastern Province

IPD SHARING:
Plan to Share IPD: No